CLINICAL TRIAL: NCT04138901
Title: Ultrasound-guided Subcostal Transversus Abdominis Plane Block in Gastric Cancer Patients Undergoing Laparoscopic Gastrectomy: A Randomized Controlled Double-blinded Study
Brief Title: Postoperative Analgesic Effect of Subcostal TAPB for Laparoscopic Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-2019-01
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Stomach neoplasms; Nerve block
MeSH Terms: conditions — Pain, Postoperative; Stomach Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: A prospective randomized double-blinded study
Who Masked: Participant, Outcomes Assessor
Masking Description: We plan to perform TAPB in patients under general anesthesia. Physicians not involved in this study will investigate the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Experimental): Patients receiving bilateral subcostal TAP block.
  Interventions: Procedure: Ultrasound guided subcostal transversus abdominis plane block (TAPB); Drug: Ropivacaine 0.75% Injectable Solution; Device: 21G 100 mm stimulator needle (Echoplex®, Vygon, Ecouen, France)
- Group C (No Intervention): Patients not receiving bilateral subcostal TAP block.

INTERVENTIONS:
Procedure: Ultrasound guided subcostal transversus abdominis plane block (TAPB) — At the end of surgery, an anesthesiologist will perform bilateral subcostal TAP block with 0.375% ropivacaine 15ml at each site under ultrasound guidance.
  Other Names: TAP block
  Arms: Group T
Drug: Ropivacaine 0.75% Injectable Solution — 0.375% ropivacaine is injected to the transversus abdominis plane via 21G 100 mm stimulator needle (Echoplex®, Vygon, Ecouen, France)
  Arms: Group T
Device: 21G 100 mm stimulator needle (Echoplex®, Vygon, Ecouen, France) — 0.375% ropivacaine is injected to the transversus abdominis plane via 21G 100 mm stimulator needle (Echoplex®, Vygon, Ecouen, France)
  Arms: Group T

SUMMARY:
This prospective, randomized, single blinded study is designed to evaluate the postoperative analgesic efficacy of the ultrasound-guided subcostal transversus abdominis plane block in gastric cancer patients undergoing laparoscopic gastrectomy. We hypothesize that US guided subcostal TAP block with ropivacaine can significantly reduce postoperative opioid comparison in patients with laparoscopic gastrectomy.

DETAILED DESCRIPTION:
Adult patients undergoing elective laparoscopic gastrectomy are randomly allocated to receive subcostal TAP block (n=56) or not (n=56), in addition to a standard postoperative analgesic regimen comprising of IV fentanyl-based patient-controlled analgesia (PCA) and NSAIDs as required. At the end of surgery, the TAP group patients will receive bilateral subcostal TAP block under ultrasound guidance with 15ml of 0.375% ropivacaine bilaterally. Each patient was assessed by a blinded investigator at 6, 12, 24, and 48 h postoperatively. The primary outcome is total fentanyl consumption at 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective laparoscopic gastrectomy under general anesthesia
* American Society of Anesthesiologists (ASA) physical classification I-III
* Consent to IV-patient controlled analgesia use
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* Do not understand our study
* Allergies to anesthetic or analgesic medications
* Wound infiltration analgesia for postoperative pain control
* Infection or anatomic abnormality at the needle insertion site
* Pregnancy/Breast feeder
* Medical or psychological disease that can affect the treatment response

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Total fentanyl consumption during 24 hours | postoperative 24 hours
  postoperative cumulative fentanyl consumption (mcg)

SECONDARY OUTCOMES:
Total fentanyl consumption | postoperative 6, 12, 48 hours
  postoperative cumulative fentanyl consumption (mcg)
Postoperative pain score | postoperative 6, 12, 24, 48 hours
  11-pointed NRS pain score at resting/coughing NRS (0-10): 0, "no pain"; 10, "worst pain imaginable"
occurrence of opioid-related side effects | postoperative 6, 12, 24, 48 hours
  Incidence of postoperative nausea and vomiting, dizziness, sedation, respiratory depression (%)
Rescue nonopioid(ketorolac, nefopam) analgesic requirement | postoperative 6, 12, 24, 48 hours
  Overall postoperative rescue of nonopoioid(ketorolac, nefopam) analgesic requirement

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No